CLINICAL TRIAL: NCT01621295
Title: Assessing the Patient Experience in Cancer Care: An Observational Communication Study
Brief Title: Assessing the Patient Experience in Cancer Care
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of Southern California (Other); Johns Hopkins University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jon C. Tilburt, PI, Mayo Clinic
Other Study IDs: 11-006682; R01AT006515 (NIH)
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Brain Neoplasm; Breast Neoplasm; Endocrine Gland Neoplasm; Gastrointestinal Neoplasm; Genitourinary Neoplasm; Gynecological Neoplasm; Head and Neck Neoplasm; Lung Neoplasm; Melanoma; Sarcoma
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Endocrine Gland Neoplasms; Gastrointestinal Neoplasms; Urogenital Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Melanoma; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Communication is an important component of comprehensive cancer care impacting patient satisfaction, adherence, and quality of life. The wide array of issues addressed in cancer clinical interactions makes communicating about a broad range of topics (including quality of life, communication, symptom control, complementary/alternative therapies, costs, treatment burden, prognosis, anxiety, side-effects, sexual function, palliative care options, etc.) especially interesting and potentially challenging. Some of these topics may not be routinely addressed in the clinical interaction or may require consultative support from other members of the comprehensive cancer care team. One frequently overlooked critical element in research on communication between cancer clinicians, their patients, and their primary care clinicians is describing real-time consultations between patients and their clinicians. These interactions provide rich material for assessing key psycho-social dynamics and identifying issues that patients find important in their care. In order to devise systems of care that optimize the patient experience, it is critical that clinicians and researchers understand, appreciate, and systematically characterize the richness and complexity of the decision-making process in routine cancer consultations between cancer patients and their treating clinicians. This study seeks to assess the patient experience in cancer care by observing patients and their physicians in their clinical interactions and following them for several months to see how their care went. By describing in-depth the conversations and experiences of patients in these clinical interactions, this study will lay the foundation for practice-based interventions to optimize patients' interactions with their cancer care teams.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Histological confirmation of: brain, breast, endocrine, gastrointestinal, genitourinary, gynecological, head/neck, lung, melanoma, or sarcoma malignancies.
* Speak English or Spanish
* Not enrolled in hospice
* In any of the following phases of the cancer control continuum: initial diagnosis, initial treatment, early survivorship, or recurrence.
* Provide written informed consent

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients age 18 or over receiving care from clinicians who have also consented to participate in this study at Mayo Clinic Rochester, University of Southern California-Norris, or LA County Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2012-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Frequency/duration/content of routine cancer consultations surrounding key topics in the clinical dialogue. | Time of enrollment through completion of 3 month follow-up survey
  Key topics to be studied include: quality of life, complementary and alternative therapies, psycho-social characteristics, patient-clinician dynamics, health literacy

CONTACTS AND LOCATIONS:
Overall Officials: Jon C Tilburt, MD, MPH, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Los Angeles County Hospital, Los Angeles, California
  - University of Southern California - Norris, Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota